CLINICAL TRIAL: NCT01381367
Title: Phase 4 Study of PPSV23 Pneumococcal Vaccine in COPD Patients Using High Daily Dose of Inhaled Corticosteroid
Brief Title: PPSV23 Pneumococcal Vaccine in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Ming-Tzer Lin, Chest Division, Department of Internal Medicine, Far Eastern Memorial Hosptial
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FEMH-97-C-037
Record Dates: First submitted 2009-02-16; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Inhaled corticosteroid; Pneumococcal vaccine; Acute exacerbation; High-dose daily inhaled corticosteroid usage; Efficacy of the PPSV23 pneumococcal vaccine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Pneumococcal Vaccines; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine (Experimental): Enrolled COPD patients receiving PPSV23 pneumococcal vaccine
  Interventions: Biological: PPSV23 pneumococcal vaccine (Pneumovax®)
- Normal saline (Placebo Comparator): Enrolled COPD patient receiving placebo normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: PPSV23 pneumococcal vaccine (Pneumovax®) — The adult anti-pneumococcal vaccine was a 23-polyvalent pneumococcal vaccine (Pneumovax®, Aventis Pastuer MSD), 0.5 ml of which was given subcutaneously. Duration of the efficacy is about 4-5 years.
  Other Names: Pneumovax®, Aventis Pastuer MSD
  Arms: Vaccine
Drug: Normal Saline — normal saline, 0.5ml given subcutaneously
  Arms: Normal saline

SUMMARY:
Streptococcus pneumoniae is the most common causes of community-acquired pneumonia and exacerbations in chronic obstructive pulmonary disease (COPD) patients, which are associated with morbidity, mortality, and higher health-care cost. In addition, recently high daily dose of inhaled corticosteroid (ICS) therapy became more evident to be beneficial in moderate-to-severe COPD patients, but excess risk of pneumonia shown in database analysis was worried about by primary physicians. The use of pneumococcal polysaccharide vaccination (PPSV23) has protective efficacy to eliminate infection of Streptococcus pneumoniae from previous studies. If the use of PPSV23 can reduce the incidence of pneumonia or exacerbations in COPD patients using high daily dose of ICS, the benefit of ICS can be preserved and risk of pneumonia can be reduced. However, there is only limited data supporting this hypothesis. In this study, the investigators will conduct a double-blinded, randomized controlled trial to evaluate the clinical efficacy of PPSV23 in severe COPD patients using high daily dose of ICS.

DETAILED DESCRIPTION:
Exacerbations are a common feature in moderate-to-severe chronic obstructive pulmonary disease (COPD). Morbidity, mortality and health-care costs of these patients largely result from exacerbations. The most common causes of an exacerbation are infection of tracheobronchial tree. Among them, Streptococcus pneumoniae is the most frequently isolated organism, accounting for 5-25% patients of COPD, while it is also the most commonly identified cause in community-acquired pneumonia (CAP), accounting for 16.5-38.9% of CAP patients.

In recent years, widespread emergence of antimicrobial resistance in Streptococcus pneumoniae has became a major global concern, especially in Taiwan, one of the highest levels of antibiotic-resistant pneumococci in the world. Therefore, primary prevention by vaccination is encouraged for those high-risk patients with COPD. The currently available adult pneumococcal vaccine consists of the capsular polysaccharide of 23 different serotypes of Streptococcus pneumoniae (PPSV23). The antibodies produced in response to this polysaccharide can provide protection by inducing host immune cells to kill or to opsonize bacteria for phagocytosis.

Until now, few studies have been designed to specifically examine vaccine efficacy in COPD patients. Among 3 available randomized controlled trials, only one study involving 596 patients found, from post-hoc analyses, some protective efficacy for pneumonia in patients of < 65 years of age and of an FEV1 < 40% predicted. Based on above evidence (only limited body of data), the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2006 Guideline has recommended the PPSV23 inoculation as evidence B.

By the way, in comparison to placebo and the single components, a superior control by means of the inhaled corticosteroids (ICS)/long-acting beta2-agonist (LABA) fixed combination therapy has been demonstrated for significant clinical improvement in moderate-to-severe COPD patients, except mortality, by meta-analysis and large prospective studies (TORCH [Towards a Revolution in COPD Health] trial and INSPIRE [Investigating New Standards for Prophylaxis in Reduction of Exacerbations] trial). However, those database indicated that high daily dose of ICS (fluticasone propionate at a dose of 500-1000mcg daily) was associated with an excess risk of pneumonia, which doubles the pneumonia incidence in patients not receiving ICS. The immunogenicity of PPSV23 in COPD patients using systemic steroid was demonstrated but the clinical efficacy of vaccination has not been investigated.

From above-mentioned background, if the use of PPSV23 can reduce the incidence of pneumonia or exacerbations in COPD patients using high daily dose of ICS, the benefit of ICS can be preserved and risk of pneumonia can be reduced. For primary physicians, this hypothesis, if true, is very beneficial. So, in this study, the investigators want to conduct a double-blinded, randomized controlled trial to evaluate the clinical efficacy of PPSV23 in COPD patients using high daily dose of ICS.

ELIGIBILITY:
Inclusion Criteria:

1. no previously vaccination with PPSV23,
2. a clinical diagnosis of severe COPD which is defined according to the GOLD 2006 guideline (11): FEV1/FVC < 70%, FEV1 reversibility test < 200 ml, and FEV1 < 50% of predicted,
3. current or past exposure of smoking,
4. no exacerbation in the month prior to enrollment,
5. age < 65 years,
6. using high daily dose of ICS (budesonide > 800-1600 mcg/day or fluticasone > 500-1000 mcg/day),
7. providing written informed consent.

Exclusion Criteria:

1. Patients are excluded from the study if they are pregnant, or have immunosuppressed status (known current neoplasm, renal insufficiency in dialysis, human immunodeficiency virus (HIV) infection, severe hepatic impairment, hypogammaglobulinemia, anatomical or functional asplenia).
2. Asthma, cystic fibrosis, bronchiectasis, and severe sequelae of pulmonary tuberculosis are also excluded by pulmonary function study and chest imaging before patient's enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
the incidence of pneumonia and exacerbations | 1 year

SECONDARY OUTCOMES:
time to the first episode of pneumonia or exacerbation | 1 year
change in lung function (post-bronchodilator FEV1, FVC) | 1 year
all cause mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Tzer Lin, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan